CLINICAL TRIAL: NCT01897532
Title: CARMELINA: A Multicenter, International, Randomized, Parallel Group, Double-blind, Placebo-controlled, Cardiovascular Safety and Renal Microvascular Outcome Study With Linagliptin, 5 mg Once Daily in Patients With Type 2 Diabetes Mellitus at High Vascular Risk
Brief Title: Cardiovascular and Renal Microvascular Outcome Study With Linagliptin in Patients With Type 2 Diabetes Mellitus (CARMELINA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.22; 2011-004148-23 (EudraCT Number)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Linagliptin (Experimental)
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — placebo matching tablets
  Arms: Placebo
Drug: Linagliptin
  Arms: Linagliptin

SUMMARY:
The aim of the study is to investigate the longterm impact on cardiovascular morbidity, mortality and renal function of treatment with linagliptin in a selected population of patients with Type 2 diabetes mellitus (T2DM) and to compare outcomes against placebo, on a background of standard of care.

ELIGIBILITY:
Inclusion criteria:

1. Documented diagnosis of T2DM before visit 1(screening).
2. Male or female patients who are drug-naïve or pre-treated with any antidiabetic background medication, excluding treatment with Glucagon-like Peptide 1 (GLP-1) receptor agonists, Dipeptidyl-peptidase 4 (DPP-4) inhibitors or Sodium Glucose Linked Transporter 2 (SGLT-2) inhibitors if => consecutive 7 days.
3. Stable antidiabetic background medication (unchanged daily dose) for at least 8 weeks prior to randomization. If insulin is part of the background therapy, the average daily insulin dose should not have changed by more than 10% within the 8 weeks prior to randomization compared with the daily insulin dose at randomization.
4. HbA1c of => 6.5% and <= 10.0% at Visit 1 (screening)
5. Age => 18 years at Visit 1(screening). For Japan only: Age => 20 years at Visit 1
6. Body Mass Index (BMI) <= 45 kg/m2 at Visit 1 (screening)
7. Signed and dated written informed consent by date of Visit 1(screening) in accordance with Good Clinical Practice (GCP) and local legislation prior to any study related procedure
8. High risk of cardiovascular (CV) events defined by: 1) albuminuria (micro or macro) and previous macrovascular disease and/or 2) impaired renal function with predefined Urine Albumin Creatinine Ratio (UACR)

Exclusion criteria:

1. Type 1 diabetes mellitus.
2. Treatment (=> 7 consecutive days) with GLP-1 receptor agonists, other DPP-4 inhibitors or SGLT-2 inhibitors prior to informed consent. Note: This also includes clinical trials where these antidiabetic drugs have been provided to the patient.
3. Active liver disease or impaired hepatic function, defined by serum levels of either Alanine Transaminase (ALT) (SGPT), Aspartate transaminase (AST) (SGOT), or alkaline phosphatase (AP) => 3 x upper limit of normal (ULN) as determined at Visit 1.
4. Estimated Glomerular filtration Rate (eGFR) <15 ml/min/1.73 m2 (severe renal impairment or End Stage Renal Disease (ESRD), Modification of Diet in Renal Disease (MDRD) formula), as determined during screening at Visit 1 and/or the need for maintenance dialysis.
5. Any previous (or planned within next 12 months) bariatric surgery (open or laparoscopic) or intervention (gastric sleeve).
6. Pre-planned coronary artery re-vascularisation (PCI, CABG) or any previous PCI and/or CABG <= 2 months prior informed consent.
7. Known hypersensitivity or allergy to the investigational products or its excipients.
8. Any previous or current alcohol or drug abuse that would interfere with trial participation in the opinion of the investigator.
9. Participation in another trial with an investigational drug ongoing or within 2 months prior to visit 1 (screening).
10. Pre-menopausal women (last menstruation = 1 year prior to informed consent) who are nursing or pregnant, are of child-bearing potential and are not practicing an acceptable method of birth control (acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence (if allowed by local authorities), double barrier method and vasectomised partner) or do not plan to continue using acceptable method of birth control throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial.
11. Patients considered unreliable by the investigator concerning the requirements for follow up during the study and/or compliance with study drug administration, have a life expectancy less than 5 years for non-CV causes, or have cancer other than non-melanoma skin cancer within last 3 years, or has any other condition than mentioned which in the opinion of the investigator, would not allow safe participation in the study.
12. Acute coronary syndrome (ACS), diagnosed <= 2 months prior to visit 1 (screening).
13. Stroke or Transient Ischemic Attack (TIA) <= 3 months prior to visit 1 (screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6991 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (645):
- United States (197):
  - Longwood Research, Huntsville, Alabama
  - Scottsboro Quick Care Clinic, Scottsboro, Alabama
  - Office of Dr. Terence T. Hart MD, Tuscumbia, Alabama
  - Arrowhead Health Centers, Glendale, Arizona
  - Precision Trials, LLC, Phoenix, Arizona
  - Harrisburg Family Medical Center, Harrisburg, Arkansas
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - Kaiser Permanente - San Diego, Bonita, Bonita, California
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Valley Research, Fresno, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Clearview Medical Research, LLC, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Office of Dr. Richard S. Cherlin, Los Gatos, California
  - Coastal Medical Research Group, Los Osos, California
  - Novo Research, Incorporated, Modesto, California
  - Providence Clinical Research, North Hollywood, California
  - Northridge Clinical Research Inc., Northridge, California
  - Carr Cardiology, Oceanside, California
  - Center for Clinical Trials of Sacramento, Incorporated, Sacramento, California
  - North America Research Institute, San Dimas, California
  - Trinitas Research, Incorporated, San Jose, California
  - Metabolic Institute of America, Tarzana, California
  - Center for Clinical Trials of San Gabriel, West Covina, California
  - Western Nephrology & Metabolic, Arvada, Colorado
  - South Denver Nephrology, Denver, Colorado
  - Colorado Center for Bone Research, P.C., Golden, Colorado
  - Helix Biomedics LLC, Boynton Beach, Florida
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Nova Clinical Research, LLC, Bradenton, Florida
  - PAB Clinical Research, Brandon, Florida
  - Meridien Research, Brooksville, Florida
  - Southeast Clinical Research, LLC, Chiefland, Florida
  - BayCare Medical Group, Clearwater, Florida
  - Cohen Medical Research Associates, LLC, Delray Beach, Florida
  - Innovation Medical Research Center, Inc, Doral, Florida
  - Integrative Research Associates, Fort Lauderdale, Florida
  - Jellinger and Lerman, MD, PA dba The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Direct Helpers Medical Center, Inc, Hialeah, Florida
  - Universal Clinical Research, Hialeah, Florida
  - Homestead Associates in Research, Homestead, Florida
  - St. Vincent's Cardiology, Jacksonville, Florida
  - Care Partners Clinical Research LLC, Jacksonville, Florida
  - Altus Research, Inc., Lake Clarke Shores, Florida
  - Meridien Research, Lakeland, Florida
  - Clinical Research of Miami, Miami, Florida
  - Prestige Clinical Research Center, Inc., Miami, Florida
  - Jesscan Medical Research, Internal Medicine, Miami, Florida
  - Clintex Research Group, Inc. Research, Miami, Florida
  - University of Miami, Miami, Florida
  - Florida Medical Center & Research Inc, Miami, Florida
  - A+ Research Incorporated, Miami, Florida
  - Unlimited Medical Research, LLC, Miami, Florida
  - Regenerate Clinical Trials, Miami, Florida
  - Sanitas Research, Miami, Florida
  - Future Care Solution, LLC, Miami, Florida
  - Research Institute of South Florida Inc, Miami, Florida
  - Tellus Clinical Research, Incorporated, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Kendall South Medical Center, Inc, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - Precision Research Organization, Miami Lakes, Florida
  - School of Clinical Research, North Miami Beach, Florida
  - Harmony Clinical Research, Incorporated, North Miami Beach, Florida
  - Magnolia Research Group, Ocala, Florida
  - Family Medical Center, Orlando, Florida
  - Peninsula Research, Inc., Ormond Beach, Florida
  - Infinity Clinical Research, LLC, Plantation, Florida
  - Intercoastal Medical Group, Endocrinology, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Professional Health Care of Pinellas, Inc., St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Laureate Clinical Research Group, LLC, Atlanta, Georgia
  - Bainbridge Medical Associates, Bainbridge, Georgia
  - Atlanta Heart Specialists, LLC, Cumming, Georgia
  - McGarity, Jr., William C., Decatur, Georgia
  - Atlanta Heart Specialists, LLC, Tucker, Georgia
  - Belleville Family Medical Associates, Ltd, Belleville, Illinois
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Chicago Clinical Research Institute, Inc., Chicago, Illinois
  - Associates in Endocrinology, Incorporated, Elgin, Illinois
  - Kidney Care Center, Nephrology, Joliet, Illinois
  - American Health Network, Avon, Indiana
  - American Health Network of Indiana, LLC, Franklin, Indiana
  - American Health Network of Indiana, LLC, Greenfield, Indiana
  - American Health Network of Indiana, LLC, Muncie, Indiana
  - Buynak Clinical Research, Valparaiso, Indiana
  - Northeast Iowa Medical Education Foundation, Waterloo, Iowa
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - Diabetes and Metabolism Associates APMC, Metairie, Louisiana
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Overlea Personal Physicians, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Delmarva Heart Research Foundation, Inc, Salisbury, Maryland
  - Endeavor Medical Research, Alpena, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - McLaren Northern Michigan Hospital, Petoskey, Michigan
  - Remedica LLC, Rochester, Michigan
  - Tri-County Research, Inc, Sterling Heights, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - Mississippi Medical Research, LLC, Carriere, Mississippi
  - Truman Medical Centers, Inc., Kansas City, Missouri
  - Kansas City Veterans Administration Medical Center, Kansas City, Missouri
  - Glacier View Cardiology, PC, Kalispell, Montana
  - Platte River Nephrology, North Platte, Nebraska
  - Omaha Veterans Affairs Medical Center, Omaha, Nebraska
  - Alas Science Clinical Research, Las Vegas, Nevada
  - USMA Clin. Research/Union Square Med. Associates, Elizabeth, New Jersey
  - Mount Sinai - PRIME, Linden, New Jersey
  - New Mexico Clinical Research and Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Life Medi-Research and Management, Brooklyn, New York
  - United Medical Associates, Johnson City, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Jacobi Medical Center, The Bronx, New York
  - Kernodle Clinic West, Burlington, North Carolina
  - Main Street Physicians Care, Calabash, North Carolina
  - Box Arthritis & Rheumatology of the Carolinas, Charlotte, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - PMG Research of Bristol, LLC, Hickory, North Carolina
  - Novant Health Southern Piedmont Primary Care, Monroe, North Carolina
  - Research Institute of the Carolinas, PLC, Mooresville, North Carolina
  - Down East Medical Associates, Morehead City, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Natalie A Doyle, M.D., P.A., Wilson, North Carolina
  - Summa Health System, Akron, Ohio
  - Medical Frontiers, LLC, Carlisle, Ohio
  - Dayton VA Medical Center, Dayton, Ohio
  - Norton Community Care, Norton, Ohio
  - Apex Medical Research, AMR, Incorporated, Springfield, Ohio
  - ProMedica Health Education & Research Corp., Toledo, Ohio
  - COR Clinical Research, LLC, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - The Corvallis Clinic, PC, Corvallis, Oregon
  - Blair Medical Associates, Altoona, Pennsylvania
  - Clinical Research Associates of Central Pennsylvania, Altoona, Pennsylvania
  - Central Bucks Cardiology, Doylestown, Pennsylvania
  - Doylestown Health Cardiology, Doylestown, Pennsylvania
  - Lycoming Internal Medicine, Inc, Jersey Shore, Pennsylvania
  - Montgomery Medical Incorporated, Smithfield, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Spectrum Medical Research, LLC, Gaffney, South Carolina
  - VitaLink Research, Greenville, South Carolina
  - Mountain View Clinical Research, Greer, South Carolina
  - Vita Link Research- Rock Hill, Rock Hill, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Holston Medical Group, Bristol, Tennessee
  - State of Franklin Healthcare Associates, PLLC, Johnson City, Tennessee
  - DCT- AACT, LLC dba Discovery Clinical Trials, Austin, Texas
  - Rockwood Medical Clinic, Bedford, Texas
  - Texas Health Physicians Group, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - The Endocrine Center, Houston, Texas
  - Texas Family Geriatrics Clinic, Houston, Texas
  - Memorial Clinical Associates Research, Houston, Texas
  - Break Through Medical Research, Irving, Texas
  - Medical & Surgical Clinic, Irving, Texas
  - West Memorial Family Practice, Katy, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - Permian Research Foundation, Odessa, Texas
  - Methodist Hospital Research Institute, Internal Medicine, Pearland, Texas
  - Health Texas Research Institute, San Antonio, Texas
  - Covenant Clinical Research, PA, San Antonio, Texas
  - DM Clinical Research, San Antonio, Texas
  - DCT-Stone Oak, LLC dba Discovery Clinical Trials, San Antonio, Texas
  - Sealy Urgent Care Center and Medical Clinic, Sealy, Texas
  - Pioneer Research Solutions, Inc., Sugar Land, Texas
  - DM Clinical Research, Tomball, Texas
  - Crossroads Clinical Research, LLC, Victoria, Texas
  - Ericksen Research & Development, LLC, Clinton, Utah
  - Focus Clinical Research, Draper, Utah
  - Advanced Research Institute, Ogden, Utah
  - Paramount Medical Care, Ogden, Utah
  - Burke Internal Medicine and Research, Burke, Virginia
  - Nova Health Management & Research Group, PC, Herndon, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - Hunter Holmes McGuire Veterans Administration Medical Center, Richmond, Virginia
  - Roanoke Heart Institute PLC, Roanoke, Virginia
  - Salem Veterans Affairs Medical Center, Salem, Virginia
  - Sound Medical Research, Port Orchard, Washington
  - Zablocki VA Medical Center, Milwaukee, Wisconsin
- Argentina (55):
  - Instituto Médico Adrogué, Adrogué
  - Hospital Interzonal General de Agudos Dr Jose Penna, Bahía Blanca
  - Inst de Inv Clinicas-Bahia Blanca, Bahía Blanca
  - Hospital Italiano Regional del Sur, Bahia Blanca, Bahía Blanca
  - Hospital Sirio-Libanés, Caba
  - Centro de Investigaciones Metabólicas, Ciudad Autonoma Buenos Aires
  - CIPREC, Ciudad Autonoma Buenos Aires
  - Hospital Italiano, Ciudad Autonoma Buenos Aires
  - Consultorios Asociados de Endocrinología e Invest Clínica, Ciudad Autonoma Buenos Aires
  - CEDIC - Centro de Investigacion Clinica, Ciudad Autonoma Buenos Aires
  - Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma Buenos Aires
  - CCBR - Buenos Aires - AR, Ciudad Autonoma Buenos Aires
  - Centro Médico Viamonte, Ciudad Autonoma de Bs As
  - Centro Universitario de Investigacion Corrientes, Corrientes
  - Centro Médico Colon, Córdoba
  - CEMAIC - Centro Medico Especializado, Córdoba
  - Inst. Privado de Inv. Clínicas de Córdoba, Córdoba
  - Sanatorio Allende S.A., Córdoba
  - Clínica Colombo, Córdoba
  - Instituto DAMIC - Fundacion Rusculleda, Córdoba
  - Hospital Cordoba, Córdoba
  - IPAC - Clínica Privada Caraffa SRL, Córdoba
  - Clinica Privada del Prado, Córdoba
  - CIPADI, Godoy Cruz
  - Centro Medico Dr. Javier Marino, Haedo
  - Hospital Italiano de La Plata, La Plata
  - Unidad de Cardiologia Clinica, Mar del Plata
  - Hospital Privado de Comunidad, Mar del Plata
  - Hospital Central de Mendoza, Mendoza, Mendoza
  - Hospital San Martin, Paraná
  - Sanatorio San Martin S.A., Venado Tuerto, Pellegrini
  - CER Instituto Médico, Quilmes
  - Instituto de Investigaciones Clínicas de Quilmes, Quilmes
  - Instituto de Investigaciones Clinicas de Rosario, Rosario
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario, Rosario
  - Instituto Medico Fundación Grupo Colaborativo Rosario, Rosario
  - Sanatorio Británico, Rosario
  - Sanatorio Norte, Rosario
  - Instituto de Hematologia y Medicina Clinica Ruben Davoli, Rosario
  - Sanatorio Delta, Rosario
  - Centro Medico CIR, Rosario
  - CEDyN, Rosario
  - Instituto CAICI, Rosario
  - Instituto Medico CENICLAR-C de Investigaciones Clinicas, Rosario
  - Centro Cardiovascular Salta, Salta
  - CORDIS S.A., Salta, Salta
  - Prevencion Cardiovascular Salta, Salta, Salta
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
  - CCBR Tucuman, San Miguel de Tucumán
  - Instituto de Investigaciones Clinicas San Nicolas, San Nicolás
  - Centro Medico Luquez, San Vicente
  - Centro de Investigaciones Clínicas del Litoral, Santa Fe
  - Hospital "Dr. José Maria Cullen ", Santa Fé
  - Clinica Privada Fusavim SRL, Villa María
  - Instituto de Investigaciones Clínicas Zárate, Zárate
- Brazil (39):
  - Hospital Universitário João de Barros Barreto, Belém
  - Hospital Felício Rocho, Belo Horizonte
  - Hospital Lifecenter, Belo Horizonte
  - Hospital Vera Cruz, Belo Horizonte
  - Hospital Angelina Caron, Campina Grande do Sul
  - HMCP - Hospital e Maternidade Celso Pierro - PUC-Campinas, Campinas
  - CAEP - Centro Avançado de Estudos e Pesquisas Ltda.,Campinas, Campinas
  - Hospital Universitário, Canoas
  - Universidade de Caxias do Sul - IPCEM - Inst. de Pesq.clilni, Caxias do Sul
  - Hospital de Caridade Santa Casa de Misericordia de Curitiba, Curitiba
  - HC UFPR, Curitiba
  - Cruz Vermelha Brasileira - Filial do Estado do Paraná, Curitiba
  - Centro de Estudos em Diabetes e Hipertensão, Fortaleza
  - Centro de Pesquisas em Diabetes e Doenças, Fortaleza
  - ICE-HUWC - Instituto Cearense de Endocrinologia, Fortaleza
  - Via Médica, Goiânia
  - Hospital Bruno Born, Lajeado
  - ICM - Instituto do Coração de Marília, Marília
  - Hospital São Vicente de Paulo, Passo Fundo
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Centro de Pesquisas em Diabetes, Porto Alegre
  - Instituto de Cardiologia Rio Grande do Sul, Porto Alegre
  - Centro de Pesquisas Médicas Básica e Clínica Ltda, Recife
  - CCBR - Rio de Janeiro - BR, Rio de Janeiro
  - Centro de Pesquisa Clínica Santa Maria, Santa Maria
  - CCBR Brasil - São Paulo, Santo André
  - Instituto Domingo Braile, São José do Rio Preto
  - Fundacao Faculdade Regional de Medicina, Sao Jose, São José do Rio Preto
  - Cpquali Pesquisa Clinica Ltda, São Paulo
  - Centro de Pesquisa Clinica - CPCLIN, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - FGM Clínica Paulista de Doenças Cardiovasculares LTDA, São Paulo
  - Hospital Sao Paulo - UNIFESP, São Paulo
  - Hospital do Servidor Público Estadual, São Paulo
  - Dr. Consulta, São Paulo
  - Hospital das Clinicas da FMUSP, São Paulo
  - Incor - Instituto do Coração - HCFMUSP, São Paulo
  - IMC - Instituto de Moléstias Cardiovasculares Tatuí, Tatuí
  - ICT - Instituto do Coração do Triângulo, Uberlândia
- Bulgaria (10):
  - MHAT - Blagoevgrad, EOOD, Blagoevgrad
  - MHAT "Yuliya Vrevska" EOOD, Byala, Byala
  - MHAT "Dr.Stambolski", Cardiology&Intensiv Care Dept,Kazanlak, Kazanlak
  - UMHAT "Kaspela", EOOD, Plovdiv, Plovdiv
  - DCC 1 - Ruse, EOOD, Rousse
  - Fifth MHAT - Sofia EAD, Sofia, Sofia
  - MHAT Lyulin, Sofia
  - MHAT 'Tokuda Hospital Sofia', EAD, Sofia
  - USHATE Hospital 'Academy Ivan Penchev', Sofia, Sofia
  - DCC "Equita" EOOD, Varna
- Canada (28):
  - ALTA Clinical Research Inc., Edmonton, Alberta
  - The Bailey Clinic, Red Deer, Alberta
  - Dr. Ronald Collette, Burnaby, British Columbia
  - The Medical Arts Health Research Group, Penticton, British Columbia
  - LMC Clinical Research dba Manna Research Inc. Vancouver, Vancouver, British Columbia
  - Fraser Clinical Trials Inc., Victoria, British Columbia
  - Discovery Clinical Services Ltd., Victoria, British Columbia
  - CookMed Research, Victoria, British Columbia
  - Winnipeg Regional Health Authority, Winnipeg, Winnipeg, Manitoba
  - True North Clinical Research Halifax, Inc., Halifax, Nova Scotia
  - LMC Endocrinology Centres (Barrie) Ltd., Barrie, Ontario
  - JBN Medical Diagnostic Services Inc., Burlington, Ontario
  - LMC Endocrinology Centres (Etobicoke) Ltd., Etobicoke, Ontario
  - Medicor Research, Greater Sudbury, Ontario
  - Sudbury Cardiac Research, Greater Sudbury, Ontario
  - Dr. R. Labonte Prof. Med. Corp, Greater Sudbury, Ontario
  - LMC Endocrinology Centres (Markham) Ltd., Markham, Ontario
  - SKDS Research Incorporated, Newmarket, Ontario
  - ViaCar Recherche Clinique Inc, Brossard, Quebec
  - Hopital Charles - LeMoyne, Greenfield Park, Quebec
  - Centre De Recherche Clinique, Laval, Quebec
  - Recherche Invascor Inc., Longueuil, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - St Jerome Medical Research Inc., Saint-Jérôme, Quebec
  - LMC Endocrinology Centres (Montreal), Saint-Laurent, Quebec
  - Recherche Clinique Sigma Inc., Québec
  - Clinique des maladies Lipidiques de Quebec, Québec
- Chile (9):
  - Hospital Regional de Punta Arenas Dr. Lautaro Navarro Avaria, Punta Arenas
  - Hospital El Pino, Santiago
  - Sociedad Medica Cardiologica El Llano, Santiago
  - Hospital Militar de Santiago, Santiago
  - Hospital Sotero del Rio, Santiago
  - CeCim - Centro de Estudios Clinicos e Investigacion Medica, Santiago
  - Hospital Padre Alberto Hurtado, Santiago
  - Hospital Base Valdivia, Valdivia
  - Hospital Naval Almirante Nef, Viña del Mar
- China (8):
  - Beijing Jishuitan Hospital, Beijing
  - Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Zhejiang University School of Medicine SIR RUN RUN SHAW Hospital, Hangzhou
  - Center Hospital of Jinan, Jinan
  - People's Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Tongji Hospital, Tongji University, Shanghai
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - General Hospital of Ningxia Medical University, Yinchuan
- Colombia (15):
  - CEQUIN, Armenia
  - Corazon IPS S.A.S., Barranquilla
  - Clínica de la Costa Ltda., Barranquilla
  - IPS Centro Cientifico Asistencia, Barranquilla
  - Centro de Atencion e Investigacion Medica S.A. - CAIMED, Bogotá
  - CAFESALUD Medicina Prepagada S.A., Bogotá
  - Dexa Diabetes Servicios Médicos Ltda, Bogotá
  - Solano y Terront Servicios Médicos Ltda., Bogotá
  - Fundacion Reina Isabel, Cali
  - IPS Centro Medico Julián Coronel S.A., Cali
  - Fundación Centro de Investigaciones Biomédicas Riescard, Espinal
  - Centro de Investigacion Clínica Avanzada, Medellín
  - Fundacion Centro de Investigacion Clinica CIC, Medellin, Medellín
  - Fundacion Centro de Obesidad y Metabolismo - COMETA, Pasto
  - Healthy Medical CenterS.A.S, Zipaquirá, Zipaquirá
- Croatia (7):
  - General Hospital Karlovac, Karlovac
  - Hospital for Medical Rehabilitation, Krapinske Toplice, Krapinske Toplice
  - General Hospital Slavonski Brod, Slavonski Brod
  - General Hospital Varazdin, Varaždin
  - General Hosp. Zadar, Dept. of Internal Medicine-Pulmonology, Zadar
  - Clinical Hospital Sveti Duh, Zagreb
  - University hospital center Zagreb, Zagreb
- Czechia (16):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Revmatologie Bruntal, s.r.o., Bruntál
  - Poliklinika Chocen, a.s., Choceň
  - Aesculap Ambulance Sro, Dolní Břežany
  - OKELI s.r.o., Hodonín
  - Nemocnice Jindrichuv Hradec a.s., Jindřichův Hradec
  - Regional Hospital Liberec, Liberec
  - InterKardioML s.r.o., Mariánské Lázně
  - Interna a diabetologicka ordinace s.r.o., Náchod
  - PreventaMed, s.r.o., Olomouc
  - Univ. Hospital Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice V Praze, Prague
  - ResTrial s.r.o., Prague
  - Thomayer Hospital, Praha 4 - Krc
  - Hospital Slany, Internal Department, Slaný
  - Krajska zdravotni, a.s. - Nemocnice Teplice, o.z., Teplice
- Germany (8):
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - Zentrum für klinische Forschung Dr. med. Irma Schöll & Kollegen, Bad Homburg
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - ClinPhenomics GmbH & Co KG, Frankfurt, Frankfurt
  - IKF Pneumologie GmbH & Co. KG, Frankfurt am Main
  - Diabetologische Schwerpunktpraxis, Hohenmölsen, Hohenmölsen
  - EUGASTRO GmbH, Leipzig, Leipzig
  - Gemeinschaftspraxis Dr. Taeschner / Dr. Bonigut, Leipzig, Leipzig
- Hungary (17):
  - Lausmed Kft. Outpatient Unit of Internal Medicine, Baja
  - Dr. Kenessey Albert Kórház-Rendelõintézet, Balassagyarmat, Balassagyarmat
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfured, Balatonfüred
  - Clinexpert Kft., Budapest
  - Obudai Egeszsegugyi Centrum, Budapest
  - QUALICLINIC Kft, Budapest
  - Semmelweis Egyetem, Budapest, Budapest
  - University Debrecen Hospital, Debrecen
  - Markhot Ferenc Hospital, Eger, Eger
  - Csongrad Megyei Eu. Ellato Kozp. Hodmezovasarhely-Mako, Hódmezővásárhely
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvar, Kaposvár
  - Selye Janos Hospital Komarom, Komárom
  - Ermellek Egeszsegcentrum, Létavértes
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klin. Kozpont, Szeged
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- Israel (10):
  - Haemek Medical Center, Afula
  - Bnei Zion Medical Center, Haifa, Haifa
  - Rambam Medical Center, Haifa
  - Herzliya Medical Center, Herzliya
  - Wolfson Medical Center, Holon
  - Hadassah Medical Center, Ein-Karem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Ziv Medical Center, Safed
  - Sourasky Medical Center, Tel Aviv
- Japan (10):
  - Daishinkai Medical Corporation Ookuma Hospital, Aichi, Nagoya
  - Seikeikai New Tokyo Heart Clinic, Chiba, Matsudo
  - Saiseikai Matsuyama Hospital, Ehime, Matsuyama
  - Aso Co.,Ltd Iizuka Hospital, Fukuoka, Iizuka
  - Kitakyushubyoin Kitakyushu General Hospital, Fukuoka, Kitakyushu
  - The Veritas Hospital, Hyogo, Kawanishi
  - Ibaraki Seinan Medical Center Hospital, Ibaraki, Sashima-gun
  - Kokan Clinic, Kanagawa, Kawasaki
  - Nagano Red Cross Hospital, Nagano, Nagano
  - Josuikai Olive Takamatsu Medical Clinic, Takamatsu
- Malaysia (10):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Tengku Ampuan Rahimah, Klang
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Monash University(Sunway Campus), Petaling Jaya
  - Hospital Pulau Pinang, Pulau Pinang
  - Universiti Putra Malaysia, Serdang
  - Hospital Seri Manjung, Seri Manjung
  - Hospital Taiping, Taiping
  - Klinik Kesihatan Tampin, Tampin
- Mexico (21):
  - Investigación en Salud y Metabolismo S.C., Chihuahua City
  - Phylasis Clinicas Research S de RL de CV, Cuautitlán Izcalli
  - Centro para el Desarrollo de la Medicina y de Asist Med Espe, Culiacán
  - Centro de Investigacion Biomedica y Farmaceutica, S.C., Distrito Federal
  - Servicios Medicos de la Pena SC, Guadalajara
  - Medical Care & Research SA de CV, Mérida
  - Sociedad de Cirugia Vascular Plastica Reconstructiva, Mérida
  - Phytomedicamenta S.A. de C.V., México
  - Comite Mexicano Para la Prevencion de Osteoporosis AC, México
  - Centro de Atención e Investigación en Factores de Riesgo, México
  - Clinstile S.A. de C.V., México
  - Ultimate Medica SA de CV, México
  - Health Pharma Professional Research S.A. de C.V., México
  - Centro de Estudios Clinicos y Especialidades Medicas, S.C., Monterrey
  - AVIX Investigación Clínica S.C, Monterrey
  - Global Trial Research Center S.A. de C.V., Monterrey
  - Centro de Investigacion Clinica Chapultepec S. A. de C. V., Morelia
  - Centro de Estudios Clínicos de Queretaro S.C., CECLIQ, Querétaro
  - Centro de Investigacion Cardiovascular y Metabolica, Tijuana
  - Centro de Investigación Médica de Ocidente, S.C., Zapopan
  - Hospital Dr Angel Leano, Zapopan
- Netherlands (10):
  - Rijnstate Hospital, Arnhem
  - Albert SchweitzerZiekenhuis, Dordrecht
  - Universitair Medisch Centrum Groningen, Groningen
  - Martini Ziekenhuis, Groningen
  - Bethesda Cardiology Group, Hoogeveen, Hoogeveen
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Rotterdam Research Institute, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
  - TweeSteden Ziekenhuis, Waalwijk
  - Gelre Ziekenhuis Zutphen, Zutphen
- Poland (32):
  - B_Serwis Popenda Sp.Jawna, Chorzów
  - Poradnia Kardiologiczna Jaroslaw Jurowiecki, Gdansk
  - University Clinical Center, Gdansk, Gdansk
  - Indywidualna Specjalistyczna Praktyka Lekarska, Gdynia
  - MCBK Iwona Czajkowska Anna Podrazka- Szczepaniak S.C., Grodzisk Mazowiecki
  - Centrum Medyczne Pratia Katowice II, Katowice
  - Polimedica Centrum Bada?, Profilaktyki I Leczenia, Kielce
  - NZOZ Centrum Medyczne ProMiMed Sp. z o.o., Sp.k., Krakow, Krakow
  - Centrum Terapii Wspolczesnej J.M., Lodz
  - CCBR - Lodz - PL, Lodz, Lodz
  - Individual Specialized Practice, Lodz
  - Centrum Medyczne "Luxmed" Sp. z o.o., Lublin
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - NZOZ Specialized Ambulance "MEDICA", Lublin
  - RCMed- Regionalne Centrum Medyczne, Nowy Duninów
  - Medicome Sp. z o.o., Oświęcim
  - Prywatny Gabinet Lekarski Lech Lazuka, Parczew
  - Clin.Hosp.Med.Univ.Marcinkowski in Poznan, Poznan
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - KOMED Marek Konieczny, Puławy
  - Indywidualna Specjalistyczna Praktyka Lekarska Dr N Med Andrzej Wittek, Ruda Śląska
  - Centrum Medyczne Medyk, Rzeszów
  - RCMed- Regionalne Centrum Medyczne, Sochaczew
  - KO-MED Centra Kliniczne Staszow, Staszów
  - NSZOZ Medicus, Środa Wielkopolska
  - Lecznice Citomed Sp. z o.o., Torun
  - NZOZ Nasz Lekarz, Torun
  - NBR Polska, Warsaw
  - CCBR/Somed - Warszaw - PL, Warsaw
  - Regionalna Poradnia Diabetoloiczna Zytkiewicz-Jaruga, Wroclaw
  - KO-MED Centra Kliniczne Zamosc, Zamość
  - Polimedica Centrum Bada?, Profilaktyki I Leczenia, Zgierz
- Portugal (7):
  - Hospital de Braga-Escala Braga, Braga
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - CHLO, EPE - Hospital S. Francisco Xavier, Lisbon
  - Hospital da Luz, Lisbon
  - Hospital CUF Porto, Porto
  - Centro Hospitalar de Vila Nova de Gaia, V. N. Gaia
- Romania (20):
  - SC Diana Barbonta SRL, Alba Iulia, Alba Iulia
  - Spitalul Universitar de Urgenta, Bucuresti, Bucharest
  - I.N.D.N.B.M. "Prof. Dr. N.C. Paulescu" - Sediul Central, Bucharest
  - CMI Dr. Stolea T. Violeta, Bucharest
  - Clinica Medicala Data Plus SRL, Bucharest
  - I.N.D.N.B.M. "Prof. Dr. N.C. Paulescu" - Sediul "I.L. Caragiale", Bucharest
  - S.C Centrul Medical "Sanatatea Ta" S.R.L, Bucharest
  - S.C. Policlinica CCBR SRL, Bucuresti, Bucharest
  - Medcon SRL, Buzău
  - Spitalul Clinic Judetean de Urgenta ¿Sf. Apostol Andrei¿, Galati
  - Spitalul Clinic, Iasi, Iași
  - Consultmed SRL, Iasi, Iași
  - SC Diaconu-Sotropa Michaela, Cabinet de Diabet, Iași
  - S.C Grandmed S.R.L, Oradea, Oradea
  - Pelican Impex SRL, Cabinet Nr. 15, Oradea
  - S.C Anamed S.R.L, Oradea
  - S.C. Diabmed Dr. Popescu Alexandrina S.R.L, Ploieşti
  - Gensan SRL, Sibiu
  - Mediab SRL, Târgu Mureş
  - Centrul Medical Dr Negrisanu SRL, Timișoara
- Russia (22):
  - SBEI HPE Altay State Medical University of MoH and SD, Barnaul
  - Res.Inst.-Compl.Iss.Cardi.Dis., Kemerovo
  - NSIH "Departmental Hospital on Station Kemerovo of OJSC "Russian Railways", Kemerovo
  - First Moscow State Medical University n.a. I.M. Sechenov, Moscow
  - Moscow 1st State Med.Univ.n.a.I.M.Sechenov, Moscow
  - SBEI HPE "Moscow State Medical and Dentistry University, Moscow
  - Moscow State Medical Dentistry University, Moscow
  - SBIH of Novosibirsk Region "Clinical Emergency Hospital #2", Novosibirsk
  - Novosibirsk Regional Clinical Cardiological Dispansary, Novosibirsk
  - FSBSI "Scientific Research Institute", Novosibirsk, Novosibirsk
  - FSBSI "Scientific and Research Institute of Physiology and Basic Medicine", Novosibirsk
  - BIH of OR "City Hospital # 2", Omsk, Omsk
  - SBIH of Perm territory " City Clinical Hospital # 2 n.a., Perm
  - SBI of Ryazan region "Regional Clinical Cardiological Dis., Ryazan
  - FSBMEI HPE "Military Medical Academy n.a. S.M. Kirov", Saint Petersburg
  - Medical Research Institute LLC, St. Petersburg, Saint Petersburg
  - 1stPavlov St.Med.Univ.St.-Petersburg Res.Inst., Saint Petersburg
  - Federal North-West Medical Research Centre, Saint Petersburg
  - SPb SBHI "City Policlinic #74", Saint Petersburg
  - SPb SBIH "City Pokrovskaya Hospital", Saint Petersburg
  - GUZ "City Clinical Hospital #40, 197706 Saint-Petersburg, Sestroretsk
  - FSBI "Research Institute for Cardiology", Tomsk
- South Africa (23):
  - Cardiology Clinical Research, Alberton
  - Iatros International, Bloemfontein
  - Limaro Research, Bloemfontein
  - Dr JM Engelbrecht Practice, Cape Town
  - Dr Dawood, Mohamed and Pillay, Cape Town
  - TREAD Research, Cape Town
  - Langeberg Clinical Trials, Cape Town
  - Cape Town Medical Research Centre, Cape Town
  - Ismail, SM, Cape Town
  - Groote Schuur Hospital, Cape Town
  - Latiff, GHVM, Durban
  - Londisizwe Research Centre, Durban, Durban
  - Diabetes Care Centre, Johannesburg
  - Wits Clinical Research Chris Hani Baragwanath Hospital, Johannesburg
  - WCR CMJAH Clinical Trial Site, Johannesburg
  - DJW Navorsing, Krugersdorp
  - Emmed Research, Pretoria
  - University of Pretoria, Pretoria
  - Syzygy Clinical Research Services, Pretoria
  - Into Research, Pretoria
  - Seeber, M, Pretoria
  - Dr M Duki Research and Trial Site, Verulam, Verulam
  - Clinical Projects Research, Worcester
- South Korea (12):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National Univ. Hosp, Busan
  - Myongji Hospital, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Wonju Severance Christian Hosp, Wŏnju
- Spain (15):
  - Hospital Virgen del Mar, Almería
  - Hospital de la Ribera, Alzira
  - Hospital Germans Trias i Pujol, Badalona
  - Specialist, Barcelona
  - CAP Sarria, Barcelona
  - Hospital Quiron. I.C.U., Barcelona
  - EBA Centelles, Centelles
  - Fundación Jiménez Díaz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital General de Segovia, Segovia
  - Hospital Quironsalud Infanta Luisa, Seville
  - Hospital Virgen Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Dr. Peset, Valencia
  - Hospital Virgen de las Montañas, Villamartin, Villamartín
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipe Veterans General Hospital, Taipei
  - Chang-Gung Memorial Hospital, Linkou, Taoyuan
- Ukraine (23):
  - Chernivtsi Regional Endocrinology Dispensary, Chernivtsi
  - Regional CH Dept of Endocrinology SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - CI Ivano-Frankivsk Reg Cl Card Center, Ivano-Frankivsk
  - L.T. Malaya Institute of Therapy AMS of Ukraine, Kharkiv
  - CIPH Prof. O.I. Meshchaninov Kharkiv CCH of A&E, Kharkiv
  - CI of Healthcare Kharkiv CCH #8, Kharkiv, Kharkiv
  - KCCC of Endocr Dept of General Endocrine Pathology, Kyiv
  - City Clinical Hospital No. 1, Kiev, Kyiv
  - V.P. Komisarenko Inst. of Endocrinology and Metabolism, Kyiv
  - Kjiv City Oleksandrivska Clinical Hospital, Kyiv
  - LLC Treatment and Diagnostic Center Adonis Plus, Kyiv, Kyiv
  - SI National Scientific Centre of Radiation Medicine of NAMSU, Kyiv
  - P.L. Shupyk NMA of PGE Ch of D H for S-ts of NASU, Kyiv
  - SI V.P.Komisarenko Institute of Endocrinology and Metabolism, Kyiv
  - Lviv Regional Endocrinology Dispensary, Lviv
  - M.V. Sklifosovskyi Poltava RCH, Poltava, Poltava
  - CI Sumy City Clinical Hospital #1 Dept of Therapy Sumy SU, Sumy
  - CI of TRC Ternopil UH, Ternopli
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - Vinnytsia RC Highly Special.Endocr.Center Dept of Therapy, Vinnytsia
  - M.I. Pyrogov VRCH, Vinnytsia, Vinnytsia
  - CCH #1 M.I. Pyrogov VNMU Ch of Propaedeutics of IM, Vinnytsia
  - CI Zapor CCH#10 SI ZMA PGE Ch of therapy clin pharmacol & endocrin, Zaporizhzhia
- United Kingdom (13):
  - University Hospital Monklands, Airdrie
  - Queen Elizabeth Hospital, Birmingham
  - Bradford on Avon Health Centre, Bradford-on-Avon
  - Ashgate Medical Practice, Chesterfield
  - Dumfries and Galloway Royal Infirmary, Dumfries
  - Ninewells Hospital & Medical School, Dundee
  - Royal Devon and Exeter Hospital, Exeter
  - Glasgow Royal Infirmary, Glasgow
  - Leicester General Hospital, Leicester
  - Barts and The London School of Medicine and Dentistry, London
  - Morriston Hospital, Swansea
  - Queen Elizabeth II Hospital, Welwyn Garden City
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Marx N, Kolkailah AA, Rosenstock J, Johansen OE, Cooper ME, Alexander JH, Toto RD, Wanner C, Espeland MA, Mattheus M, Schnaidt S, Perkovic V, Gollop ND, McGuire DK. Hypoglycemia and Cardiovascular Outcomes in the CARMELINA and CAROLINA Trials of Linagliptin: A Secondary Analysis of Randomized Clinical Trials. JAMA Cardiol. 2024 Feb 1;9(2):134-143. doi: 10.1001/jamacardio.2023.4602. PMID 38170502
- [Derived] Balasubramanian P, Kernan WN, Sheth KN, Ofstad AP, Rosenstock J, Wanner C, Zinman B, Mattheus M, Marx N, Inzucchi SE. Baseline Cardiovascular Risk Factor Control in Patients With Type 2 Diabetes and Coronary Disease Versus Stroke: Secondary Analysis of Cardiovascular Outcome Trials. Stroke. 2023 Aug;54(8):2013-2021. doi: 10.1161/STROKEAHA.122.042053. Epub 2023 Jul 14. PMID 37449424
- [Derived] Dar MS, Wanner C, Marx N, Ofstad AP, Mattheus M, Kaspers S, Beg SA. Cardiovascular outcomes trial data from EMPA-REG OUTCOME, CAROLINA and CARMELINA: Assessment of a novel staging system for type 2 diabetes. Diabetes Obes Metab. 2023 May;25(5):1372-1384. doi: 10.1111/dom.14989. Epub 2023 Mar 6. PMID 36700391
- [Derived] Verhagen C, Janssen J, Minderhoud CA, van den Berg E, Wanner C, Passera A, Johansen OE, Biessels GJ. Chronic kidney disease and cognitive decline in patients with type 2 diabetes at elevated cardiovascular risk. J Diabetes Complications. 2022 Oct;36(10):108303. doi: 10.1016/j.jdiacomp.2022.108303. Epub 2022 Aug 31. PMID 36116359
- [Derived] Verhagen C, Janssen J, Exalto LG, van den Berg E, Johansen OE, Biessels GJ. Diabetes-specific dementia risk score (DSDRS) predicts cognitive performance in patients with type 2 diabetes at high cardio-renal risk. J Diabetes Complications. 2020 Oct;34(10):107674. doi: 10.1016/j.jdiacomp.2020.107674. Epub 2020 Jul 16. PMID 32723590
- [Derived] Perkovic V, Toto R, Cooper ME, Mann JFE, Rosenstock J, McGuire DK, Kahn SE, Marx N, Alexander JH, Zinman B, Pfarr E, Schnaidt S, Meinicke T, von Eynatten M, George JT, Johansen OE, Wanner C; CARMELINA investigators. Effects of Linagliptin on Cardiovascular and Kidney Outcomes in People With Normal and Reduced Kidney Function: Secondary Analysis of the CARMELINA Randomized Trial. Diabetes Care. 2020 Aug;43(8):1803-1812. doi: 10.2337/dc20-0279. Epub 2020 May 22. PMID 32444457
- [Derived] Biessels GJ, Verhagen C, Janssen J, van den Berg E, Zinman B, Rosenstock J, George JT, Passera A, Schnaidt S, Johansen OE; CARMELINA Investigators. Effect of Linagliptin on Cognitive Performance in Patients With Type 2 Diabetes and Cardiorenal Comorbidities: The CARMELINA Randomized Trial. Diabetes Care. 2019 Oct;42(10):1930-1938. doi: 10.2337/dc19-0783. Epub 2019 Aug 9. PMID 31399442
- [Derived] McGuire DK, Alexander JH, Johansen OE, Perkovic V, Rosenstock J, Cooper ME, Wanner C, Kahn SE, Toto RD, Zinman B, Baanstra D, Pfarr E, Schnaidt S, Meinicke T, George JT, von Eynatten M, Marx N; CARMELINA Investigators. Linagliptin Effects on Heart Failure and Related Outcomes in Individuals With Type 2 Diabetes Mellitus at High Cardiovascular and Renal Risk in CARMELINA. Circulation. 2019 Jan 15;139(3):351-361. doi: 10.1161/CIRCULATIONAHA.118.038352. PMID 30586723
- [Derived] Rosenstock J, Perkovic V, Johansen OE, Cooper ME, Kahn SE, Marx N, Alexander JH, Pencina M, Toto RD, Wanner C, Zinman B, Woerle HJ, Baanstra D, Pfarr E, Schnaidt S, Meinicke T, George JT, von Eynatten M, McGuire DK; CARMELINA Investigators. Effect of Linagliptin vs Placebo on Major Cardiovascular Events in Adults With Type 2 Diabetes and High Cardiovascular and Renal Risk: The CARMELINA Randomized Clinical Trial. JAMA. 2019 Jan 1;321(1):69-79. doi: 10.1001/jama.2018.18269. PMID 30418475
- [Derived] Rosenstock J, Perkovic V, Alexander JH, Cooper ME, Marx N, Pencina MJ, Toto RD, Wanner C, Zinman B, Baanstra D, Pfarr E, Mattheus M, Broedl UC, Woerle HJ, George JT, von Eynatten M, McGuire DK; CARMELINA(R) investigators. Rationale, design, and baseline characteristics of the CArdiovascular safety and Renal Microvascular outcomE study with LINAgliptin (CARMELINA(R)): a randomized, double-blind, placebo-controlled clinical trial in patients with type 2 diabetes and high cardio-renal risk. Cardiovasc Diabetol. 2018 Mar 14;17(1):39. doi: 10.1186/s12933-018-0682-3. PMID 29540217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to initiation of any trial-related procedure, all patients were informed about the trial verbally and in writing by the investigator. The patients signed and dated the informed consent before any study related procedures.
Pre-assignment Details: Patients with documented diagnosis of Type 2 Diabetes Mellitus (T2DM) at high risk of cardiovascular (CV) events and who met all the inclusion criteria and did not meet any of the exclusion criteria could be enrolled in the trial.
Groups:
- Placebo: Patients were administered Placebo matching Linagliptin 5 mg film-coated tablet orally once daily.
  At Visit 2, patients received one treatment box sufficient for 12 weeks treatment (plus 1 week reserve).
  At Visit 3 (until trial end) patients received 2 medication boxes sufficient for 24 weeks treatment (plus 2 weeks reserve).
- Linagliptin: Patients were administered Linagliptin 5 milligram (mg) film-coated tablet orally once daily.
  At Visit 2, patients received one treatment box sufficient for 12 weeks treatment (plus 1 week reserve).
  At Visit 3 (until trial end) patients received 2 medication boxes sufficient for 24 weeks treatment (plus 2 weeks reserve).
Period: Discontinuation From Treatment
Arm/Group | Placebo | Linagliptin
Started (Randomised) | 3492 | 3499
Treated | 3485 | 3494
Completed (Not prematurely discontinued from trial medication) | 2530 | 2660
Not Completed | 962 | 839
Not completed — Not Treated | 7 | 5
Not completed — Other reason than specified | 196 | 176
Not completed — Withdrawal by Subject | 333 | 281
Not completed — Non compliance | 24 | 15
Not completed — Adverse event/ CV outcome event | 402 | 362
Period: Discontinuation From Trial
Arm/Group | Placebo | Linagliptin
Started (Randomised) | 3492 | 3499
Treated | 3485 | 3494
Completed (Completed the trial or died) | 3430 | 3458
Not Completed | 62 | 41
Not completed — Not Treated | 7 | 5
Not completed — Patient lost to follow-up for MACE | 55 | 36

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All patients treated with at least one dose of trial medication. If no trial medication was taken at site during the visit, but the medication kit was dispensed to the patient and not all trial medication was returned, the patient was included in the TS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin | Total
Number analyzed (Participants) | 3485 | 3494 | 6979
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (9.14) | 66.1 (9.05) | 65.9 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1243 | 1346 | 2589
  Male | 2242 | 2148 | 4390
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1274 | 1227 | 2501
  Not Hispanic or Latino | 2211 | 2267 | 4478
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 156 | 159 | 315
  Asian | 333 | 307 | 640
  Native Hawaiian or Other Pacific Islander | 10 | 7 | 17
  Black or African American | 217 | 194 | 411
  White | 2769 | 2827 | 5596
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Occurrence of Any of the Following Adjudication-confirmed Components of the Primary Composite Endpoint 3-point Major Adverse Cardiovascular (CV) Events (3-point MACE): CV Death, Non-fatal Myocardial Infarction (MI) or Non-fatal Stroke.
Description: Time to event analysis of patients with first occurrence of any of the following adjudication-confirmed components of the primary composite endpoint (3-point MACE): CV death, non-fatal MI or non-fatal stroke. The percentage of observed patients with first occurrence of any of the following adjudication-confirmed components of the primary composite endpoint (3-point MACE) was reported.
Time Frame: From randomization to individual end of observation; up to 4.3 years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 3485 | 3494
percentage of participants | 12.1 | 12.4
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Cox proportional hazard regression model was performed to compare the effect of linagliptin versus placebo. Model included randomised treatment and geographical region as factors. Breslow's method was used for dealing with ties. First hypothesis (non-inferiority of the primary endpoint) was to be tested at the one-sided alpha-level of 2.5%. In case of significance the next set of hypotheses (two separate hypothesis tests) were to be tested with a sequentially rejective multiple test procedure; Test type: Non-Inferiority — The non-inferiority margin was chosen as 1.3 (FDA Guidance for Industry - Diabetes Mellitus - Evaluating Cardiovascular Risk in New Antidiabetic Therapies to Treat Type 2 Diabetes); p = 0.0002, Regression, Cox — p-value for Hazard ratio (HR) ≥1.3 (1-sided); Based on a Cox regression model with terms for treatment group and region; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.89 to 1.17]
Statistical Analysis 2: Comparison: Placebo vs Linagliptin; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.6301, Regression, Cox — p-value for HR ≥1.0 (1-sided); Based on a Cox regression model with terms for treatment group and region; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.89 to 1.17]

2. Secondary Outcome: Time to the First Occurrence of Any of the Following Adjudication-confirmed Components: Renal Death, Sustained End Stage Renal Disease (ESRD), or Sustained Decrease of 40% or More in Estimated Glomerular Filtration Rate (eGFR).
Description: Time to the first occurrence of any of the following adjudication-confirmed components: renal death, sustained ESRD, or sustained decrease of 40% or more in eGFR.
  The percentage of observed patients with first occurrence of any of the following adjudication-confirmed components: renal death, sustained ESRD, or sustained decrease of 40% or more in eGFR was reported.
Time Frame: From randomization to individual end of observation; up to 4.3 years
Population: TS
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 3485 | 3494
percentage of participants | 8.8 | 9.4
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.6918, Regression, Cox — p-value for HR ≥1.0 (1-sided); Based on a Cox regression model with terms for treatment group and region; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.89 to 1.22]

ADVERSE EVENTS:
Time Frame: Adverse events with an onset after the first dose of trial medication up to a period of 7 days after the last permanent study drug stop; up to 4.3 years
Arm/Group | Placebo | Linagliptin
All-Cause Mortality (participants affected / at risk) | 253/3485 | 250/3494
Serious Adverse Events (participants affected / at risk) | 1343/3485 | 1293/3494
Other Adverse Events (participants affected / at risk) | 1422/3485 | 1434/3494
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3485) | Linagliptin (N=3494)
Pneumonia (Infections and infestations) | 121 | 99
Urinary tract infection (Infections and infestations) | 41 | 30
Cellulitis (Infections and infestations) | 38 | 22
Sepsis (Infections and infestations) | 33 | 18
Bronchitis (Infections and infestations) | 17 | 8
Osteomyelitis (Infections and infestations) | 14 | 11
Septic shock (Infections and infestations) | 12 | 13
Gangrene (Infections and infestations) | 14 | 10
Gastroenteritis (Infections and infestations) | 9 | 11
Localised infection (Infections and infestations) | 7 | 10
Pyelonephritis (Infections and infestations) | 3 | 14
Urosepsis (Infections and infestations) | 7 | 5
Respiratory tract infection (Infections and infestations) | 7 | 3
Diabetic foot infection (Infections and infestations) | 6 | 3
Influenza (Infections and infestations) | 2 | 7
Pyelonephritis acute (Infections and infestations) | 3 | 6
Erysipelas (Infections and infestations) | 4 | 3
Infected skin ulcer (Infections and infestations) | 6 | 1
Lower respiratory tract infection (Infections and infestations) | 4 | 3
Abscess limb (Infections and infestations) | 4 | 2
Device related infection (Infections and infestations) | 2 | 4
Peritonitis (Infections and infestations) | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Bacteraemia (Infections and infestations) | 2 | 3
Necrotising fasciitis (Infections and infestations) | 3 | 2
Postoperative wound infection (Infections and infestations) | 2 | 3
Anal abscess (Infections and infestations) | 4 | 0
Catheter site infection (Infections and infestations) | 3 | 1
Diabetic gangrene (Infections and infestations) | 3 | 1
Diverticulitis (Infections and infestations) | 2 | 2
Lung infection (Infections and infestations) | 1 | 3
Post procedural infection (Infections and infestations) | 3 | 1
Subcutaneous abscess (Infections and infestations) | 4 | 0
Appendicitis (Infections and infestations) | 3 | 0
Arthritis bacterial (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 2
Endocarditis (Infections and infestations) | 2 | 1
Escherichia sepsis (Infections and infestations) | 1 | 2
Infection (Infections and infestations) | 1 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 2
Pulmonary sepsis (Infections and infestations) | 1 | 2
Soft tissue infection (Infections and infestations) | 1 | 2
Bacterial infection (Infections and infestations) | 1 | 1
Carbuncle (Infections and infestations) | 1 | 1
Cholecystitis infective (Infections and infestations) | 2 | 0
Device related sepsis (Infections and infestations) | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 2
Intervertebral discitis (Infections and infestations) | 0 | 2
Osteomyelitis chronic (Infections and infestations) | 1 | 1
Paronychia (Infections and infestations) | 2 | 0
Periodontitis (Infections and infestations) | 2 | 0
Scrotal abscess (Infections and infestations) | 0 | 2
Staphylococcal infection (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 2 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Blebitis (Infections and infestations) | 1 | 0
Bursitis infective (Infections and infestations) | 1 | 0
Chikungunya virus infection (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Clostridium colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Fungal peritonitis (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Gastroenteritis shigella (Infections and infestations) | 1 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
H1n1 influenza (Infections and infestations) | 0 | 1
Hepatitis c (Infections and infestations) | 1 | 0
Hepatitis infectious mononucleosis (Infections and infestations) | 1 | 0
Histoplasmosis cutaneous (Infections and infestations) | 1 | 0
Histoplasmosis disseminated (Infections and infestations) | 0 | 1
Infected cyst (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1
Infectious colitis (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Injection site abscess (Infections and infestations) | 0 | 1
Intestinal sepsis (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0
Leptospirosis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Lyme disease (Infections and infestations) | 1 | 0
Mediastinitis (Infections and infestations) | 1 | 0
Medical device site cellulitis (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 1
Mycoplasma infection (Infections and infestations) | 0 | 1
Myiasis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Nosocomial infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis viral (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pneumonia chlamydial (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Pulpitis dental (Infections and infestations) | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Scrub typhus (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Spinal cord abscess (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Systemic infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Viraemia (Infections and infestations) | 0 | 1
Viral tonsillitis (Infections and infestations) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 14
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 9
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 8
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoma in situ of penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chest wall tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mucinous cystadenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Naevoid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sebaceous adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour of ampulla of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 17 | 19
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 2
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2
Drug hypersensitivity (Immune system disorders) | 0 | 1
Overlap syndrome (Immune system disorders) | 1 | 0
Goitre (Endocrine disorders) | 2 | 2
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Adrenal mass (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 38 | 28
Hyperkalaemia (Metabolism and nutrition disorders) | 19 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 22 | 12
Dehydration (Metabolism and nutrition disorders) | 6 | 11
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 10 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 7 | 9
Fluid overload (Metabolism and nutrition disorders) | 11 | 5
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 5 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 6
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 7
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 | 3
Electrolyte imbalance (Metabolism and nutrition disorders) | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4
Gout (Metabolism and nutrition disorders) | 1 | 2
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 3 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 2
Fluid retention (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1
Acquired mixed hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Fluid imbalance (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperosmolar state (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 | 1
Delirium (Psychiatric disorders) | 4 | 4
Major depression (Psychiatric disorders) | 3 | 2
Mental status changes (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Hallucination, visual (Psychiatric disorders) | 2 | 0
Acute stress disorder (Psychiatric disorders) | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 1
Affect lability (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Drug use disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Mood disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 49 | 61
Syncope (Nervous system disorders) | 25 | 15
Transient ischaemic attack (Nervous system disorders) | 9 | 27
Cerebrovascular accident (Nervous system disorders) | 12 | 10
Haemorrhagic stroke (Nervous system disorders) | 8 | 10
Dementia (Nervous system disorders) | 6 | 8
Diabetic neuropathy (Nervous system disorders) | 5 | 7
Seizure (Nervous system disorders) | 6 | 5
Cerebral infarction (Nervous system disorders) | 8 | 2
Presyncope (Nervous system disorders) | 7 | 2
Carotid artery stenosis (Nervous system disorders) | 6 | 2
Cerebral ischaemia (Nervous system disorders) | 4 | 2
Facial paralysis (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 4 | 1
Loss of consciousness (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 0 | 4
Encephalopathy (Nervous system disorders) | 2 | 2
Haemorrhage intracranial (Nervous system disorders) | 1 | 3
Hemiparesis (Nervous system disorders) | 4 | 0
Myelopathy (Nervous system disorders) | 3 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 2
Diabetic coma (Nervous system disorders) | 1 | 2
Epilepsy (Nervous system disorders) | 2 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 2
Lacunar infarction (Nervous system disorders) | 2 | 1
Basal ganglia infarction (Nervous system disorders) | 2 | 0
Brain oedema (Nervous system disorders) | 1 | 1
Brain stem infarction (Nervous system disorders) | 1 | 1
Carotid artery occlusion (Nervous system disorders) | 2 | 0
Cerebrovascular disorder (Nervous system disorders) | 2 | 0
Dementia with lewy bodies (Nervous system disorders) | 2 | 0
Embolic stroke (Nervous system disorders) | 1 | 1
Facial nerve disorder (Nervous system disorders) | 1 | 1
Hemiplegia (Nervous system disorders) | 0 | 2
Hypoglycaemic coma (Nervous system disorders) | 1 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 2
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Parkinson's disease (Nervous system disorders) | 1 | 1
Partial seizures (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 0 | 2
Thrombotic stroke (Nervous system disorders) | 1 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 1
Brain injury (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Carotid artery dissection (Nervous system disorders) | 1 | 0
Carotid sinus syndrome (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Incoherent (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Lacunar stroke (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 0 | 1
Myasthenia gravis (Nervous system disorders) | 1 | 0
Neuritis cranial (Nervous system disorders) | 0 | 1
Neuroglycopenia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Post stroke seizure (Nervous system disorders) | 0 | 1
Spinal claudication (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Spinal epidural haematoma (Nervous system disorders) | 0 | 1
Thalamic infarction (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Uraemic encephalopathy (Nervous system disorders) | 1 | 0
Vascular headache (Nervous system disorders) | 1 | 0
Vith nerve paralysis (Nervous system disorders) | 1 | 0
Wernicke's encephalopathy (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 13 | 11
Glaucoma (Eye disorders) | 9 | 6
Vitreous haemorrhage (Eye disorders) | 5 | 6
Retinal detachment (Eye disorders) | 5 | 4
Diabetic retinopathy (Eye disorders) | 4 | 3
Macular hole (Eye disorders) | 2 | 4
Retinal vein occlusion (Eye disorders) | 1 | 3
Ulcerative keratitis (Eye disorders) | 2 | 2
Diplopia (Eye disorders) | 2 | 1
Macular degeneration (Eye disorders) | 2 | 1
Angle closure glaucoma (Eye disorders) | 1 | 1
Macular fibrosis (Eye disorders) | 1 | 1
Neovascular age-related macular degeneration (Eye disorders) | 2 | 0
Retinal haemorrhage (Eye disorders) | 2 | 0
Acquired corneal dystrophy (Eye disorders) | 1 | 0
Amaurosis (Eye disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 0 | 1
Cataract cortical (Eye disorders) | 0 | 1
Corneal decompensation (Eye disorders) | 0 | 1
Cystoid macular oedema (Eye disorders) | 0 | 1
Diabetic retinal oedema (Eye disorders) | 0 | 1
Dry age-related macular degeneration (Eye disorders) | 0 | 1
Hyalosis asteroid (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 0 | 1
Open angle glaucoma (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal artery embolism (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 1
Retinal degeneration (Eye disorders) | 1 | 0
Retinopathy (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Vitreous haematoma (Eye disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 3 | 4
Vertigo (Ear and labyrinth disorders) | 4 | 3
Deafness (Ear and labyrinth disorders) | 2 | 1
Deafness bilateral (Ear and labyrinth disorders) | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 0 | 2
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Conductive deafness (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 104 | 104
Cardiac failure congestive (Cardiac disorders) | 98 | 77
Angina unstable (Cardiac disorders) | 70 | 77
Acute myocardial infarction (Cardiac disorders) | 59 | 78
Myocardial infarction (Cardiac disorders) | 54 | 47
Angina pectoris (Cardiac disorders) | 25 | 42
Atrial fibrillation (Cardiac disorders) | 26 | 34
Coronary artery disease (Cardiac disorders) | 21 | 26
Cardiac failure chronic (Cardiac disorders) | 20 | 24
Cardiac arrest (Cardiac disorders) | 17 | 25
Myocardial ischaemia (Cardiac disorders) | 12 | 20
Acute coronary syndrome (Cardiac disorders) | 18 | 12
Left ventricular failure (Cardiac disorders) | 12 | 13
Atrial flutter (Cardiac disorders) | 11 | 13
Cardiogenic shock (Cardiac disorders) | 12 | 8
Atrioventricular block complete (Cardiac disorders) | 10 | 9
Cardiac failure acute (Cardiac disorders) | 7 | 10
Cardio-respiratory arrest (Cardiac disorders) | 8 | 8
Coronary artery stenosis (Cardiac disorders) | 8 | 5
Bradycardia (Cardiac disorders) | 6 | 5
Sinus node dysfunction (Cardiac disorders) | 4 | 7
Acute left ventricular failure (Cardiac disorders) | 8 | 1
Atrioventricular block second degree (Cardiac disorders) | 4 | 5
Coronary artery occlusion (Cardiac disorders) | 3 | 6
Arteriosclerosis coronary artery (Cardiac disorders) | 6 | 2
Atrioventricular block (Cardiac disorders) | 5 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 3 | 4
Ventricular tachycardia (Cardiac disorders) | 3 | 3
Cardiomyopathy (Cardiac disorders) | 2 | 2
Cardiopulmonary failure (Cardiac disorders) | 1 | 3
Ventricular fibrillation (Cardiac disorders) | 3 | 1
Arrhythmia (Cardiac disorders) | 1 | 2
Cardiovascular insufficiency (Cardiac disorders) | 1 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 2 | 1
Ventricular arrhythmia (Cardiac disorders) | 3 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 1
Bundle branch block left (Cardiac disorders) | 1 | 1
Cardiac disorder (Cardiac disorders) | 0 | 2
Cardiomegaly (Cardiac disorders) | 2 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 2
Myocardial fibrosis (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 2
Silent myocardial infarction (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1
Systolic dysfunction (Cardiac disorders) | 1 | 1
Adams-stokes syndrome (Cardiac disorders) | 1 | 0
Aortic valve disease (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiomyopathy acute (Cardiac disorders) | 1 | 0
Cardiorenal syndrome (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Chordae tendinae rupture (Cardiac disorders) | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 1
Degenerative mitral valve disease (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial necrosis (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Paroxysmal atrioventricular block (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Sinus arrest (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Trifascicular block (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Hypertension (Vascular disorders) | 18 | 32
Hypertensive crisis (Vascular disorders) | 20 | 16
Peripheral arterial occlusive disease (Vascular disorders) | 17 | 18
Deep vein thrombosis (Vascular disorders) | 14 | 12
Peripheral artery occlusion (Vascular disorders) | 12 | 5
Peripheral ischaemia (Vascular disorders) | 11 | 5
Aortic stenosis (Vascular disorders) | 5 | 8
Peripheral vascular disorder (Vascular disorders) | 7 | 6
Extremity necrosis (Vascular disorders) | 9 | 3
Hypotension (Vascular disorders) | 7 | 5
Peripheral artery stenosis (Vascular disorders) | 4 | 3
Orthostatic hypotension (Vascular disorders) | 0 | 6
Aortic aneurysm (Vascular disorders) | 1 | 4
Hypovolaemic shock (Vascular disorders) | 1 | 4
Venous thrombosis limb (Vascular disorders) | 2 | 3
Arteriosclerosis (Vascular disorders) | 3 | 1
Hypertensive emergency (Vascular disorders) | 2 | 2
Circulatory collapse (Vascular disorders) | 1 | 2
Accelerated hypertension (Vascular disorders) | 1 | 1
Angiopathy (Vascular disorders) | 1 | 1
Diabetic macroangiopathy (Vascular disorders) | 2 | 0
Dry gangrene (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 2 | 0
Intermittent claudication (Vascular disorders) | 0 | 2
Peripheral embolism (Vascular disorders) | 2 | 0
Thrombophlebitis (Vascular disorders) | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 2
Varicose ulceration (Vascular disorders) | 0 | 2
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0
Arterial insufficiency (Vascular disorders) | 0 | 1
Arterial rupture (Vascular disorders) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1
Diabetic vascular disorder (Vascular disorders) | 0 | 1
Distributive shock (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Embolism arterial (Vascular disorders) | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 1
Orthostatic hypertension (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1
Systolic hypertension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Vascular insufficiency (Vascular disorders) | 1 | 0
Vein rupture (Vascular disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 28 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 16
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 13 | 16
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 15 | 13
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 14 | 12
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mendelson's syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paraneoplastic pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Portopulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 | 9
Gastritis (Gastrointestinal disorders) | 8 | 5
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 8
Diarrhoea (Gastrointestinal disorders) | 2 | 9
Abdominal pain (Gastrointestinal disorders) | 5 | 5
Pancreatitis acute (Gastrointestinal disorders) | 3 | 7
Inguinal hernia (Gastrointestinal disorders) | 5 | 4
Pancreatitis (Gastrointestinal disorders) | 3 | 6
Vomiting (Gastrointestinal disorders) | 3 | 6
Constipation (Gastrointestinal disorders) | 4 | 4
Pancreatitis chronic (Gastrointestinal disorders) | 6 | 2
Abdominal hernia (Gastrointestinal disorders) | 5 | 2
Large intestine polyp (Gastrointestinal disorders) | 3 | 4
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 4
Intestinal obstruction (Gastrointestinal disorders) | 3 | 3
Colitis ischaemic (Gastrointestinal disorders) | 1 | 4
Gastric ulcer (Gastrointestinal disorders) | 2 | 3
Chronic gastritis (Gastrointestinal disorders) | 1 | 3
Haematochezia (Gastrointestinal disorders) | 2 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Duodenal ulcer (Gastrointestinal disorders) | 3 | 0
Duodenitis (Gastrointestinal disorders) | 3 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Hiatus hernia (Gastrointestinal disorders) | 2 | 1
Melaena (Gastrointestinal disorders) | 0 | 3
Pancreatic cyst (Gastrointestinal disorders) | 3 | 0
Umbilical hernia (Gastrointestinal disorders) | 3 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Anal polyp (Gastrointestinal disorders) | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal vascular ectasia (Gastrointestinal disorders) | 0 | 1
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Intestinal polyp (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Mesenteric haemorrhage (Gastrointestinal disorders) | 1 | 0
Oedema mouth (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatic failure (Gastrointestinal disorders) | 0 | 1
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Retroperitoneal fibrosis (Gastrointestinal disorders) | 0 | 1
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 1
Vomiting projectile (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 9 | 10
Cholecystitis acute (Hepatobiliary disorders) | 7 | 10
Cholecystitis (Hepatobiliary disorders) | 3 | 7
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 5
Hepatic failure (Hepatobiliary disorders) | 2 | 3
Bile duct stone (Hepatobiliary disorders) | 2 | 2
Biliary colic (Hepatobiliary disorders) | 0 | 2
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Biliary dyspepsia (Hepatobiliary disorders) | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 24 | 21
Skin ulcer (Skin and subcutaneous tissue disorders) | 10 | 7
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 2
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ichthyosis acquired (Skin and subcutaneous tissue disorders) | 0 | 1
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 1
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 17 | 15
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 3
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Diabetic arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Periostitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 100 | 96
End stage renal disease (Renal and urinary disorders) | 45 | 38
Chronic kidney disease (Renal and urinary disorders) | 32 | 49
Renal failure (Renal and urinary disorders) | 31 | 32
Renal impairment (Renal and urinary disorders) | 27 | 24
Diabetic nephropathy (Renal and urinary disorders) | 7 | 9
Nephrolithiasis (Renal and urinary disorders) | 7 | 5
Urinary retention (Renal and urinary disorders) | 6 | 5
Haematuria (Renal and urinary disorders) | 4 | 5
Nephrotic syndrome (Renal and urinary disorders) | 2 | 7
Azotaemia (Renal and urinary disorders) | 6 | 1
Nephropathy (Renal and urinary disorders) | 4 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 4
Ureterolithiasis (Renal and urinary disorders) | 1 | 4
Urinary tract obstruction (Renal and urinary disorders) | 2 | 2
Calculus bladder (Renal and urinary disorders) | 0 | 2
Nephropathy toxic (Renal and urinary disorders) | 1 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 1
Renal mass (Renal and urinary disorders) | 1 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 1
Hypertensive nephropathy (Renal and urinary disorders) | 1 | 0
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal pain (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 8 | 4
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 2
Uterine polyp (Reproductive system and breast disorders) | 2 | 0
Acquired phimosis (Reproductive system and breast disorders) | 0 | 1
Cervical polyp (Reproductive system and breast disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal leukoplakia (Reproductive system and breast disorders) | 1 | 0
Accessory spleen (Congenital, familial and genetic disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Cystic lymphangioma (Congenital, familial and genetic disorders) | 1 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 1 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0
Keratosis follicular (Congenital, familial and genetic disorders) | 1 | 0
Myocardial bridging (Congenital, familial and genetic disorders) | 0 | 1
Death (General disorders) | 23 | 16
Non-cardiac chest pain (General disorders) | 15 | 15
Sudden death (General disorders) | 20 | 10
Cardiac death (General disorders) | 5 | 7
Asthenia (General disorders) | 8 | 2
Chest pain (General disorders) | 4 | 3
Pyrexia (General disorders) | 2 | 5
Multiple organ dysfunction syndrome (General disorders) | 2 | 3
Generalised oedema (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 3 | 1
Sudden cardiac death (General disorders) | 3 | 1
Chest discomfort (General disorders) | 1 | 2
Vascular stent restenosis (General disorders) | 1 | 2
Catheter site haemorrhage (General disorders) | 0 | 2
Chills (General disorders) | 0 | 2
Complication associated with device (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 0 | 2
Necrobiosis (General disorders) | 0 | 2
Application site haemorrhage (General disorders) | 0 | 1
Chronic fatigue syndrome (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Feeling abnormal (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Injection site haematoma (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Medical device site joint inflammation (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Strangulated hernia (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 1
Vascular stent occlusion (General disorders) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 30 | 36
Lipase increased (Investigations) | 5 | 4
Blood creatinine increased (Investigations) | 3 | 1
Blood pressure increased (Investigations) | 1 | 2
Arteriogram coronary (Investigations) | 0 | 2
Blood glucose increased (Investigations) | 0 | 2
Glycosylated haemoglobin increased (Investigations) | 2 | 0
Troponin increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Aspiration bronchial (Investigations) | 1 | 0
Catheterisation cardiac (Investigations) | 0 | 1
Creatinine renal clearance decreased (Investigations) | 1 | 0
Echocardiogram (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram qt prolonged (Investigations) | 1 | 0
Electrocardiogram t wave inversion (Investigations) | 0 | 1
Influenza a virus test positive (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Intracardiac pressure increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 0 | 1
Prostatic specific antigen increased (Investigations) | 1 | 0
Staphylococcus test positive (Investigations) | 1 | 0
Urine output decreased (Investigations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 25 | 19
Femur fracture (Injury, poisoning and procedural complications) | 6 | 10
Hip fracture (Injury, poisoning and procedural complications) | 7 | 3
Limb injury (Injury, poisoning and procedural complications) | 5 | 5
Road traffic accident (Injury, poisoning and procedural complications) | 7 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 5
Tibia fracture (Injury, poisoning and procedural complications) | 3 | 4
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 3
Rib fracture (Injury, poisoning and procedural complications) | 1 | 5
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 5
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 2
Head injury (Injury, poisoning and procedural complications) | 3 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 3 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 2
Patella fracture (Injury, poisoning and procedural complications) | 1 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 3 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 2
Overdose (Injury, poisoning and procedural complications) | 2 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 3 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1
Hyphaema (Injury, poisoning and procedural complications) | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 1 | 0
Colon injury (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Heart injury (Injury, poisoning and procedural complications) | 1 | 0
Incomplete spinal fusion (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Postoperative delirium (Injury, poisoning and procedural complications) | 0 | 1
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Scar (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Stoma site polyp (Injury, poisoning and procedural complications) | 1 | 0
Stomal hernia (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Vith nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Coronary revascularisation (Surgical and medical procedures) | 1 | 2
Hospitalisation (Surgical and medical procedures) | 0 | 1
Peripheral endarterectomy (Surgical and medical procedures) | 1 | 0
Homicide (Social circumstances) | 0 | 1
Limb prosthesis user (Social circumstances) | 0 | 1
Device malfunction (Product Issues) | 2 | 2
Device failure (Product Issues) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3485) | Linagliptin (N=3494)
Urinary tract infection (Infections and infestations) | 162 | 196
Hypoglycaemia (Metabolism and nutrition disorders) | 1003 | 1022
Hyperglycaemia (Metabolism and nutrition disorders) | 240 | 208
Hypertension (Vascular disorders) | 232 | 216
Glomerular filtration rate decreased (Investigations) | 200 | 202

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT01897532/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT01897532/SAP_001.pdf